CLINICAL TRIAL: NCT04903418
Title: Assessment of Relationship Between Maxillary Sinus Floor and Maxillary Posterior Teeth Root Tips Position in a Sample of Egyptian Population Using CBCT: An Observational Cross-Sectional Study
Brief Title: Assessment of Relationship Between Maxillary Sinus Floor and Maxillary Posterior Teeth Root Tips Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Tarek Khater Mohamed, Principal Investigator, Cairo University
Other Study IDs: MSF-Max. Post. teeth root tips
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CBCT software — * Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.
  * All the CBCT examinations will be obtained for patients who were scanned using CBCT Software (Planmeca Romexis® Viewer software).
  * CBCT images will be analysed in different planes.

SUMMARY:
There have been no cross-sectional studies conducted on the Egyptian population studying the relationship between maxillary sinus floor and the maxillary posterior root tips position using CBCT, and whether the maxillary sinus mucosal thickening is associated with periapical lesions as well as periodontal disease. Such study will raise the diagnostic and interpretational abilities of dental radiologists and decision making of oral surgeons and endodontists.

DETAILED DESCRIPTION:
II-Introduction In the human body, the first and largest, sinus to develop is the Maxillary Sinus (MS). The growth of this sinus begins in the intrauterine period of life, and reaches its maximum size and forms the shape of a pyramid by the time of the third molar eruption or at the age of approximately 21 years. The inferior wall of sinus is lined with Schneiderian membrane which is the unique lining of the nasal cavity and paranasal sinuses (Kilic et al., 2010). Normally, the thickness of the Schneiderian membrane is approximately 1 mm (Cakur B et al., 2013; Borgonovo et al., 2015).

Odontogenic sinusitis is the most common result of iatrogenic injury of Schneiderian membrane which could result in its thickening due to inflammatory reaction (Troeltzsch et al., 2015; Zirk et al., 2017). Tooth extraction, posterior maxillary dental implant placement, sinus lift, and orthognathic surgery are the main cause relations of odontogenic sinusitis. Other potential causes include periodontal and periapical diseases (Pen˜arrocha-Oltra et al., 2020).

Detailed study of the proximity of the maxillary posterior teeth root apices to the maxillary sinus floor (MSF) is a mandatory step before some procedures as endodontic procedures in order to avoid over-instrumentation or over-filling of restorative materials. Pushing foreign material into the MS may result in the spread of infection (Obayashiet al., 2004).

The condition of maxillary posterior teeth is usually examined by periapical and panoramic radiographs during routine dental visits. However, plain films are 2-dimensional to represent the 3-dimensional structures which make it difficult to evaluate the actual relation between sinus floor and adjacent teeth (Whyte et al., 2019).

Computed tomography (CT) is considered the gold standard for sinus diagnosis (Mafee et al., 2006). However, recently, cone beam computed tomography (CBCT) is widely utilized in oral and maxillofacial region and provides several advantages over traditional CT, including lower radiation dose and chair side process (Scarfe et al., 2006).

The use of CBCT to assess the presence and possible spread of infection from the periapical area to the MSF achieved prompt radiological diagnosis and allowed superior treatment options and minimized the possibility of complications (Oberli et al., 2007; Estrela et al., 2008; Nunes et al., 2016).

Several 3-D radiographic studies involving the maxillofacial region revealed apical protrusion of the maxillary root apices into the MS but with significant variation between populations (Mudgade, D. K. et al., 2018; Hameed, K. S. et al., 2020) Considering the individual variations of position between different maxillary posterior teeth, the aim of this study is to detect the relationship between maxillary sinus floor and the maxillary posterior root tips position, and to find the association between periapical lesions as well as periodontal disease and maxillary sinus mucosal thickening in a sample of Egyptian population using cone-beam computed tomography (CBCT).

6c. Specific objectives: To detect the relationship between maxillary sinus floor and root tips position of maxillary premolars versus maxillary molars

To find the association between periapical lesions and maxillary sinus mucosal thickening

To find the association between periodontal disease and maxillary sinus mucosal thickening

Hypothesis: null

Statement of the Problem Close relationship of maxillary posterior teeth root tips to maxillary sinus may lead to perforation of its floor, formation of oro-antral fistula, or root displacement into the maxillary sinus during endodontic treatment, tooth extraction, or any surgical procedure. Other conditions, including, periapical infection and periodontal diseases may have a precursor effect on the occurrence of sinus mucosal thickening. Therefore, accurate evaluation of the anatomic relationship of maxillary sinus and posterior teeth is crucial in the clinical practice for preoperative treatment planning in order to avoid such complications.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans for patients aged from 20 to 70 years.
* CBCT scans for patients with at least first and second maxillary premolars and first and secon maxillary molars present on one side (fully erupted teeth and fully formed apices).
* CBCT scans taken for pre-evaluation of endodontic treatment, implant placement, impacted teeth removal, obstructive sleep apnea treatment, pre-orthodontic or pre-prosthetic evaluation.
* Good quality CBCT scans.

Exclusion Criteria:

* CBCT scans for patients with no maxillary posterior teeth.
* CBCT scans for patients with history of maxillary sinus operation (including sinus floor elevation).
* CBCT scans for patients with sign or history of non-odontogenic sinusitis, including air-fluid level, thickening of all the sinus walls and maxillary sinus polyps.
* CBCT scans for patients with syndromes, congenital or developmental anomalies.
* CBCT scans for patients with bone disease.
* CBCT scans for patients with traumatic injuries to the maxillofacial region.
* Low quality CBCT scans (any artifact).

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The CBCT data of this study will be obtained from the CBCT data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt. Being a retrospective study, CBCT scans of Egyptian patients who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning will be included according to the proposed eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
using CBCT software in measurement the Relationship between maxillary sinus floor and root tips position of maxillary premolars versus maxillary molars | through study completion, an average of 1 year
  Numerical data (quantitative data)

SECONDARY OUTCOMES:
The association between presence of periapical lesions and maxillary sinus mucosal thickening | through study completion, an average of 1 year
  Categorical nominal data (percent)

OTHER OUTCOMES:
The association between presence of periodontal disease and maxillary sinus mucosal thickening | through study completion, an average of 1 year
  Categorical nominal data (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Dina F Abdelrahim, Ass. Prof., Study Director — Associate Professor Department of Oral and Maxillofacial Radiology Faculty of Dentistry